CLINICAL TRIAL: NCT03017742
Title: A Multi-Center Study on the Utility of Non-invasive Carboxyhemoglobin and Total Hemoglobin Measurement in Emergency Department Patients
Brief Title: Utility of Non-invasive Carboxyhemoglobin and Total Hemoglobin Measurement in the Emergency Department
Status: Terminated | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SUNE0002
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Results first posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-06

CONDITIONS: Carbon Monoxide Poisoning; Anemia
MeSH Terms: conditions — Carbon Monoxide Poisoning; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Test Group (Experimental): The subjects enrolled in the test group will receive the pulse oximeter
  Interventions: Device: Pulse Oximeter

INTERVENTIONS:
Device: Pulse Oximeter

SUMMARY:
The purpose of this study is to determine the clinical utility of triage screening for anemia and carbon monoxide poisoning (COP) in the ED setting.This is a prospective, nonrandomized, multi-center study of the performance of simultaneous non-invasive testing for two common disorders (COP and anemia). We will determine the limits of agreement and performance characteristics of non-invasive carboxyhemoglobin (SpCO) and hemoglobin (SpHb) values compared to standard blood tests for measurement of carboxyhemoglobin and hemoglobin, in the emergency department setting.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 year or older.
* At least one digit has acceptable width as measured by study-provided digit gauge.
* Presenting to emergency department for any complaint.
* Potential for IV catheter and/or blood draw for CBC as standard of care.

Exclusion Criteria:

* Patients unable to consent for any reason
* Patients with fingernail polish, discoloration or trauma to fingers

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 813 (Actual)
Dates: Start 2016-11; Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tepecik Training and Research Hospital IEC, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Group: The subjects enrolled in the test group will receive the pulse oximeter for various physiological parameters
Period: Overall Study
Arm/Group | Test Group
Started | 813
Completed | 740
Not Completed | 73
Not completed — Protocol Violation | 36
Not completed — Withdrawal by Subject | 37

BASELINE CHARACTERISTICS:
Groups:
- Test Group: The subjects enrolled in the test group will receive the pulse oximeter
  Pulse Oximeter
Arm/Group | Test Group
Number analyzed (Participants) | 740
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 52
  Between 18 and 65 years | 559
  >=65 years | 129
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 399
  Male | 341
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 740

OUTCOME MEASURES:

1. Primary Outcome: Difference Between SpCO and COHb
Description: Measure the difference between noninvasive carboxyhemoglobin (SpCO) and carboxyhemoglobin determined by co-oximeter measurement of blood (COHb) as calculated in terms of standard deviation.
  The average difference between paired Masimo noninvasive carboxyhemoglobin (SpCO) and reference carboxyhemoglobin (COHb) determined by co-oximeter measurement of blood represented as mean bias.
Time Frame: Up to 3 hours
Population: 140 subjects excluded due to: 35 subjects: no valid reference COHb measurements available 17 subjects: no SpCO measurements available 65 subjects: COHb sample more than 10 minutes from the SpCO measurement. 22 subjects: low SpCO confidence value
  1 subject: invalid reference measurement (COHb) Target subject sample size of 3000 was not met to evaluate difference between SpCO and COHb. The results are reported in terms of standard deviation.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Test Group
Number analyzed (Participants) | 600
percent | 2.01 (2.49)

2. Primary Outcome: SpCO Detection of Carbon Monoxide Poisoning (COP)
Description: Diagnostics performance of SpCO for detecting COP measured by sensitivity and specificity compared to COHb.
Time Frame: up to 3 hours
Population: Out of the 600 subjects that were analyzed from all that were enrolled, only 26 subjects met the criteria for carbon monoxide poisoning.
Measure: Number; unit: percentage
Arm/Group | Test Group
Number analyzed (Participants) | 600
percentage
  Sensitivity of COP Detection | 73.08
  Specificity of COP Detection | 82.75

3. Primary Outcome: Utility of SpCO as a Screening Tool for Carbon Monoxide Poisoning
Description: Surveying healthcare providers whether SpCO screening lead to identification of occult toxicity
Time Frame: up to 3 hours
Population: Clinician survey were not conducted or collected to perform data analysis.
Arm/Group | Test Group
Number analyzed (Participants) | 0

4. Primary Outcome: Carbon Monoxide (CO) Elimination Pharmacokinetics in Relation to Oxygen Administration
Description: CO elimination will be evaluated as a function of administered oxygen.
Time Frame: up to 3 hours
Population: No COHb elimination pharmacokinetics data was collected.
Arm/Group | Test Group
Number analyzed (Participants) | 0

5. Primary Outcome: Specificity of SpHb in Detecting Anemia.
Description: Specificity in detecting true non-anemic subjects as determined by co-oximeter reference analyzer.
Time Frame: up to 3 hours
Population: Excluded subjects are shown below:
  20 subjects: no valid blood reference results 73 subjects: time between the first valid SpHb reading and the venous blood draw exceeded 10 minutes.
  32 subjects: low Perfusion Index quality. 3 subjects: low signal stability 26 subjects: low SpHb confidence 18 subjects : no SpHb result displayed. 21 subjects: user error
  1 subject: pregnant
Measure: Number; unit: percentage of true negative
Arm/Group | Test Group
Number analyzed (Participants) | 546
percentage of true negative | 81.00

6. Primary Outcome: Sensitivity of SpHb Detection of Anemia.
Description: Sensitivity in detecting true anemic subjects as determined by co-oximeter reference analyzer.
Time Frame: up to 3 hours
Population: as for outcome 5
Measure: Number; unit: percent of true positives
Arm/Group | Test Group
Number analyzed (Participants) | 546
percent of true positives | 60.77

7. Primary Outcome: SpHb Utility for Screening Anemia
Description: Establish SpHb threshold that predicts the clinical outcome for acute treatment of anemia
Time Frame: up to 3 hours
Population: The number of subjects requirement defined by the study protocol were not met in this study, thus the threshold that predicts the outcome of "acute treatment of anemia" cannot be determined nor validated.
Arm/Group | Test Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout study duration, which was up to three hours.
Arm/Group | Test Group
All-Cause Mortality (participants affected / at risk) | 0/813
Serious Adverse Events (participants affected / at risk) | 0/813
Other Adverse Events (participants affected / at risk) | 0/813

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT03017742/Prot_SAP_000.pdf